CLINICAL TRIAL: NCT00692848
Title: The Impact of Procalcitonin on the Management of Children Aged 1 to 36 Month Presenting With a Fever Without a Source
Brief Title: Impact of Procalcitonin on the Management of Children Aged 1 to 36 Month Presenting With a Fever Without a Source
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Sergio Manzano MD, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: URG73
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Procalcitonin; Fever Without Source; Bacterial Infection; Bacteremia
Keywords: Procalcitonin; Antibiotic; Fever without source; Fever without focus; bacteremia; Urinary tract infection
MeSH Terms: conditions — Bacterial Infections; Bacteremia; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCT+ (Experimental): Investigations include CBC, blood culture, urine analysis and culture and procalcitonin. In this arm procalcitonin result is revealed to the attending physician. The decision to treat with antibiotics or to hospitalize was left to him
  Interventions: Other: Procalcitonin dosage PCT-Q test (Brahms, Germany)
- PCT- (No Intervention): Investigations include CBC, blood culture, urine analysis and culture and procalcitonin. In this arm, procalcitonin is not revealed to the attending physician. The decision to treat with antibiotics or to hospitalize was left to him.

INTERVENTIONS:
Other: Procalcitonin dosage PCT-Q test (Brahms, Germany) — Procalcitonin result available to the attending physician
  Other Names: PCT-Q test (Brahms, Germany)
  Arms: PCT+

SUMMARY:
Serious bacterial infections are often difficult to detect in children with fever without source. Procalcitonin is a better blood marker of infection than White blood cell count and possibly than C-reactive protein. This could lead to a reduction in antibiotic prescription. Our objective is to evaluate the impact of Procalcitonin result on antibiotic prescription in children 1 to 36 month old with fever without source and our hypothesis is that it will lower the antibiotic prescription rate

ELIGIBILITY:
Inclusion Criteria:

* Children 1-36 months
* With rectal temperature >38.0 C
* And no identified source of infection after history and physical examination

Exclusion Criteria:

* acquired or congenital immunodeficiency

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Difference in prescription of antibiotics between the two groups, excluding those treated for a bacterial infection identified by the ED investigations

SECONDARY OUTCOMES:
Difference in hospitalization rate between the two groups (excluding those hospitalized for an identified infection)
Procalcitonin sensitivity and specificity

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Manzano, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine Emergency Department, Montreal, Quebec, Canada